## Insul-In This Together Program: Optimizing Familybased Interventions for Adolescents With Type 1 Diabetes and Their Parents

Statistical Analysis Plan
NCT04589689
May 11, 2021

## Statistical Analysis Plan

- 1. Planned sample size was 150 enrolled parent-adolescent dyads. The final sample included 157 parent-adolescent dyads.
- 2. <u>Basic two-sided t-tests</u> for primary and secondary outcomes using a p-value cutoff of <.05. Compared participants based on condition assignments: intervention versus waitlisted control.
- 3. <u>Simple regression models</u>: test main effects on outcomes at 3-month and 6-month follow-ups (in Mplus)
  - a. Covariates: Teen age, diabetes duration, baseline TIR, baseline QOL, and baseline outcome (if other than TIR or QOL)
  - b. Auxiliary variables (to inform data imputation, but not directly included in model): Teen gender, baseline A1c, Teen PAID, and Parent PAID
- 4. <u>Moderation analyses</u>: separate regression models for each outcome that include set of covariates and an interaction term of condition x moderator.
  - a. Covariates: age, diabetes duration, baseline QOL, and baseline TIR
  - b. Outcomes: QOL, TIR, A1c, Teen PAID, and Parent Paid
  - c. Moderators (at baseline):
    - 1. Closed loop
    - 2. A1c  $\leq 7.5\%$
    - 3. TIR  $\geq 70\%$
    - 4. Race/ethnicity
    - 5. Income
    - 6. Insurance
    - 7. Baseline level of corresponding outcome
- 5. Mediation analyses: single mediator models
  - a. Mediator: immediate posttest
  - b. Outcomes: 3-month and 6-month follow-ups
- 6. <u>12-month follow-up</u> combine both conditions and look through 6-months (but for control the 6-month value 12-month value)



## **Moderation Models**



